CLINICAL TRIAL: NCT02375516
Title: Drug Abuse Prevention Programming for Hispanic Adolescents
Brief Title: Preventing Drug Abuse Among Hispanic Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AAAK6105; R01DA031477 (NIH)
Record Dates: First submitted 2014-02-25; First posted 2015-03-02 (Estimated); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Drug Abuse
Keywords: Drug abuse
MeSH Terms: conditions — Substance-Related Disorders | interventions — National Program of Cancer Registries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prevention Program (Experimental): Youths in the intervention-arm will interact online with the initial intervention program between pretest and posttest measurement occasions and will interact with booster sessions subsequent to 1- and 2-year follow-up measurement occasions.
  Interventions: Behavioral: Prevention Program
- Control group (No Intervention): Youths assigned to the control arm will receive no intervention.

INTERVENTIONS:
Behavioral: Prevention Program — Youths in the intervention-arm will interact online with the initial intervention program between pretest and posttest measurement occasions and will interact with booster sessions subsequent to 1- and 2-year follow-up measurement occasions. Owing to the expense associated with developing a treatment-as-usual intervention for computer delivery in the control arm, youths assigned to the control arm will receive no intervention.
  Arms: Prevention Program

SUMMARY:
The planned research aims to delay the onset of drug use and reduce harmful use and abuse among Hispanic youths. The culturally-tailored prevention program will be delivered to youths by computer. Over 5 years, the program will be developed and tested in a randomized clinical trial. The intervention program will include 10 initial sessions, followed by annual booster sessions. Outcome measurements will involve baseline, post-intervention, and three annual follow-up data collections.

The study's primary hypothesis is that rates of 30-day alcohol and drug use will be lower among participants assigned to receive the intervention. If proven to be efficacious, the program will be revised and disseminated nationally.

DETAILED DESCRIPTION:
America's largest ethnic minority group, Hispanics are also a youthful population: one-third of Hispanic Americans are less than 18 years old. Unfortunately, young Hispanic Americans are an at-risk population more likely than their majority culture peers to drop out of school, become involved in the criminal justice system, fall prey to violence, and face lifelong economic problems. Hispanic youths are also at risk for early drug use and subsequent harmful use and abuse. As early as eighth grade and relative to their Black and White peers, Hispanic adolescents report higher rates of most harmful substances. Drug use continues to pose problems for Hispanic youths throughout adolescence and into adulthood.

ELIGIBILITY:
Inclusion Criteria:

* 12 to 15 years old
* Hispanic ethnicity

Exclusion Criteria:

* None

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 678 (Actual)
Dates: Start 2012-09; Primary Completion 2019-07-01 (Actual); Study Completion 2021-04-07 (Actual)

PRIMARY OUTCOMES:
Change in average number of drug abuse instances | Baseline, Post-intervention, Year 1, Year 2, Year 3
  Measures will ask participants to report, for the past 30 days, the number of: drinks of alcohol consumed, cigarettes smoked, puffs of marijuana, and times they consumed five or more drinks during one drinking occasion. Participants will also report past 30-day use of: inhalants, ecstasy, club drugs, prescription drugs for recreational use, heroin, diet pills, and hallucinogens.

CONTACTS AND LOCATIONS:
Overall Officials: Traci Schwinn, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Schinke SP, Schwinn TM, Hursh HA. Preventing Drug Abuse Among Hispanic Adolescents: Developing a Responsive Intervention Approach. Res Soc Work Pract. 2015 Oct;25(7):794-800. doi: 10.1177/1049731514538103. Epub 2014 Jul 1. PMID 26500421
- [Result] Schwinn TM, Schinke SP, Hopkins J, Thom B. Risk and protective factors associated with adolescent girls' substance use: Data from a nationwide Facebook sample. Subst Abus. 2016 Oct-Dec;37(4):564-570. doi: 10.1080/08897077.2016.1154495. Epub 2016 Sep 20. PMID 27648525